CLINICAL TRIAL: NCT06313528
Title: A Randomized, Double-Blind, Phase 1 Study to Investigate the Effect of LY3437943 Versus Placebo on Calorie Intake and Energy Expenditure in Participants With Obesity Under Calorie Restriction
Brief Title: A Study to Measure Calorie Consumption and Usage in Participants With Obesity Using LY3437943
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18726; J1I-MC-GZBW (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-03-11; First posted 2024-03-15 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: Food; Diet
MeSH Terms: conditions — Obesity | interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3437943 (Experimental): LY3437943 administered subcutaneously (SC)
  Interventions: Drug: LY3437943
- Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LY3437943 — Administered SC
  Arms: LY3437943
Other: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of the study is to look at the effect of the study drug compared to placebo on calorie intake, energy metabolism, and appetite. The study will last up to 6 months and may include up to 20 visits.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than 30 kg/m2
* History of at least 1 self-reported unsuccessful dietary effort to reduce body weight

Exclusion Criteria:

* Change in body weight of greater than 5 kg (11 pounds) within 3 months prior to start of study
* Any of the following treatments for obesity within 1 year prior, or plan to undergo any of these during the study period: liposuction, cryolipolysis, or abdominoplasty
* Prior or planned bariatric or gastric sleeve surgery, endoscopic therapy, or device-based therapy for obesity
* Type 1 or Type 2 Diabetes, history of ketoacidosis, or hyperosmolar state
* Family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome Type 2
* Acute or chronic hepatitis
* Had within 90 days prior: acute myocardial infarction, cerebrovascular accident (stroke), coronary artery revascularization, hospitalization for unstable angina, or hospitalization due to congestive heart failure
* History of active or unstable major depressive disorder or other severe psychiatric disorder within 2 years prior
* History of chronic or acute pancreatitis
* Blood transfusion or severe blood loss within the last 3 months or hemoglobinopathy, hemolytic anemia, sickle cell anemia
* Clinically significant multiple or severe drug allergies
* Started treatment with or changed dose within 12 months prior any medications that are associated with significant weight gain
* History of substance use disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Total Calorie Intake at Lunch and Dinner (Combined) | Baseline up to Week 17 (inclusive)

SECONDARY OUTCOMES:
Change from Baseline in Sleep Metabolic Rate (SMR) | Baseline up to Week 16 (inclusive)
  In participants who achieve target weight loss
Change from Baseline in SMR | Baseline up to Week 16 (inclusive)
Change from Baseline in 24-hour Energy Expenditure (EE) | Baseline up to Week 16 (inclusive)
  In participants who achieve target weight loss
Change from Baseline in 24-hour EE | Baseline up to Week 16 (inclusive)
Change from Baseline in Total Calorie Intake at Lunch | Baseline up to Week 17 (inclusive)
Change from Baseline in Total Calorie Intake at Dinner | Baseline up to Week 17 (inclusive)
Change from Baseline in Fasting Appetite Visual Analog Score (VAS) | Baseline up to Week 16 (inclusive)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - AdventHealth Orlando, Orlando, Florida
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Measure Calorie Consumption and Usage in Participants With Obesity Using LY3437943 — https://trials.lilly.com/en-US/trial/468355